CLINICAL TRIAL: NCT05451862
Title: Holmium-166 Transarterial Radioembolization in Unresectable, Early Stage Hepatocellular Carcinoma; a Prospective, Single-arm, Open Label, Multicenter Phase II Study: HOMIE-166.
Brief Title: Holmium-166 Transarterial Radioembolization in Unresectable, Early Stage Hepatocellular Carcinoma.
Acronym: HOMIE-166
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The HOMIE-166 clinical investigation was prematurely terminated due to sponsor's decision to permanently stop production of QuiremSpheres™ and QuiremScouts™.
Sponsor: Terumo Europe N.V. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T142E3
Record Dates: First submitted 2022-06-30; First posted 2022-07-11 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Hepatocellular Carcinoma
Keywords: early stage HCC; TARE; SIRT; radioembolization; Holmium-166
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 166Ho-TARE treatment (Other): Patients with unresectable HCC with a single nodule ≤ 8 cm or up to three nodules with a diameter of ≤ 5 cm (each). Those patients who fulfil the initial selection criteria will undergo a work-up procedure for further screening of 166Ho-TARE eligibility. If a patient is deemed eligible for 166Ho-TARE, the patient will be included in the study.
  Interventions: Device: Holmium-166 treatment; Device: Holmium-166 work-up

INTERVENTIONS:
Device: Holmium-166 treatment — Implantation into hepatic tumors by delivery via the hepatic artery for the treatment of unresectable HCC liver tumors.
  Other Names: QuiremSpheresTM Holmium-166 Microspheres
Device: Holmium-166 work-up — Evaluation of lung-shunt, extrahepatic deposition and intrahepatic distribution of intra-arterially injected microspheres for patients that are eligible for TARE treatment.
  Other Names: QuiremScoutTM Holmium-166 Microspheres

SUMMARY:
166Ho-TARE is a promising modality for the treatment of HCC, given the unique characteristics of holmium, allowing careful patient selection and personalized dosimetry treatment planning. Further clinical evidence is needed to evaluate the safety and efficacy of 166Ho-TARE in the treatment of HCC patients with limited tumor burden, well preserved liver function and performance status and ineligible for liver transplantation and/or liver resection. This study will also provide further evidence on the dose-response relationship of 166Ho-TARE in (early) HCC.

DETAILED DESCRIPTION:
This is a prospective, single-arm, open-label, multicenter study with 166Ho-TARE in unresectable HCC patients with limited tumor burden and well-preserved liver function and performance status, ineligible for liver transplantation and/or liver resection. Eligibility for liver transplantation and liver resection is determined by the multidisciplinary tumor board. However, patients eligible for liver transplantation can still be included in the setting of bridge to transplant.

The study proposes to use 166Ho-TARE, including both therapeutic 166Ho-microspheres (QuiremSpheres™ Holmium-166 Microspheres) and scout 166Ho-microspheres (QuiremScout™ Holmium-166 Microspheres). All patients providing informed consent and meeting the selection criteria will be further screened using a scout dose of 166Ho-microspheres to evaluate 166Ho-TARE eligibility. Patients not eligible for selective 166Ho-TARE are considered screen failures and will not be considered as enrolled.

The primary endpoint will be assessed by blinded, independent central review, organized by an imaging core laboratory.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Multidisciplinary tumor board decision for locoregional treatment
3. Freely given, written informed consent
4. Patients with unresectable HCC with a single nodule ≤ 8 cm or up to three nodules with a diameter of ≤ 5 cm (each) eligible for selective radioembolization (including position changes of infusion catheters)
5. Non-cirrhotic patients or Child-Pugh A cirrhosis
6. ECOG performance status 0-1
7. Using an acceptable method of contraception throughout the study until survival follow up (for subjects of childbearing potential)
8. Adequate hematological, renal and liver function.

Adequate hematological function defined as:

* Hemoglobin ≥ 6 mmol/L (9.7 g/dL)
* WBC ≥ 3.0 x 10E9/L
* Absolute neutrophil count ≥ 1.5 x 10E9/L
* Platelet count ≥ 50,000/mm3

Adequate renal function defined as:

* Serum urea and serum creatinine < 1.5 times upper limit of normal (ULN)
* Creatinine clearance ≥ 45 ml/min

Adequate liver function defined as:

* Total bilirubin ≤ 35µmol/L (2.05 mg/dL)
* Albumin ≥ 30 g/L
* AST and ALT ≤ 5X ULN

Exclusion Criteria:

1. Diffuse and/or infiltrative HCC (defined as HCC consisting of multiple tiny liver nodules spreading throughout the entire liver or entire lobe, without a dominant nodule)
2. Hypoperfused HCC (defined as a lack of tumor blush (i.e. reduced or no uptake of contrast fluid) observed on the intra-procedural CT)
3. No full, selective arterial coverage on intra-procedural CT
4. Life expectancy < 6 months
5. Child-Pugh score ≥7 points
6. Prior liver transplantation
7. Prior locoregional or systemic anti-cancer therapy for HCC and previous malignancies
8. Macrovascular invasion (defined as macrovascular invasion of the hepatic and/or portal vein main branches)
9. Extrahepatic metastases
10. Clinically significant ascites
11. Hepatic encephalopathy
12. Untreated active hepatitis B and/or C
13. Work-up imaging showing:

    * Lung shunt > 30 Gy is simulated on 166Ho-scout imaging; or
    * Uncorrectable extrahepatic deposition of simulated 166Ho-scout dose activity. Activity in the falciform ligament, portal lymph nodes and gallbladder is accepted; or
    * Anticipated ineffective tumor targeting (< 150 Gy mean tumor simulated absorbed dose) of 166Ho-scout for each lesion; or
    * Entire tumor burden not within the perfused liver volume (possible extrahepatic collateral supply of the tumor); or
    * Perfused liver volume > 50% of whole liver tissue
14. Pregnant or breast-feeding
15. Current or history of cancer other than HCC, except adequately treated non-melanoma skin cancer or carcinoma in situ of the cervix
16. In the Investigator's opinion there is a reason that could limit the patient's ability to participate in the study, compliance with follow-up requirements or impact the scientific integrity of the study
17. Concurrently enrolled in another study, unless it is an observational non-interventional study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2023-08-21 (Actual); Primary Completion 2025-05-27 (Actual); Study Completion 2025-05-27 (Actual)

PRIMARY OUTCOMES:
confirmed Objective Response Rate (ORR) by localized mRECIST | 5 years
  ORR is defined as the proportion of patients achieving either complete or partial tumor response during the study, as assessed by blinded central image review according to localized mRECIST

SECONDARY OUTCOMES:
Best ORR based on localized mRECIST | 5 years
  The number and percent of patients with a confirmed response
Best and confirmed ORR based on mRECIST | 5 years
  The number and percent of patients with a confirmed response
Duration of Response (DoR) ≥ 6 months based on localized mRECIST and mRECIST | 5 years
  The number and percent of patients with a DoR ≥ 6 months. DoR is measured from time of initial response until radiological progression. Radiological progression is determined by blinded central image review according to localized mRECIST and mRECIST.
Time to Progression (TTP) | 5 years
  TTP defined as the time from treatment with QuiremSpheresTM Holmium-166 Microspheres to progression as per mRECIST
Progression-Free Survival (PFS) | 5 years
  PFS defined as the time from treatment with QuiremSpheresTM Holmium-166 Microspheres to the date of radiological progression or death from any cause. Radiological progression is determined by blinded central image review according to mRECIST
hepatic Progression-Free Survival (hPFS) | 5 years
  hPFS defined as the time from treatment with QuiremSpheresTM Holmium-166 Microspheres to the date of radiological progression in the liver or death from any cause. Radiological progression is determined by blinded central image review according to mRECIST
Liver transplantation rate | 5 years
  The number and percent of patients receiving a liver transplant
Liver resection rate | 5 years
  The number and percent of patients undergoing a liver resection
Overall survival (OS) | 5 years
  The median overall survival time
Safety and toxicity by evaluating the number of adverse events and the number of patients with each event | 5 years
  Adverse events classified by Common Terminology Criteria for Adverse Events (CTCAE) v5.0. (including clinical and laboratory toxicity)
Liver function during follow-up ALBI score | 5 years
  ALBI score
Liver function during follow-up using MELD score | 5 years
  MELD score
Liver function during follow-up using Child Pugh score | 5 years
  Child Pugh score
Assessment of dosimetry and biodistribution based on quantitative assessment of imaging scans | 5 years
  Correlation between scout and treatment for extrahepatic dose deposition, including lung shunt and digestive shunting of QuiremSpheresTM Holmium-166 Microspheres.
Assessment of dosimetry and biodistribution based on quantitative assessment of imaging scans | 5 years
  Correlation between treatment-based absorbed dose (into the tumor and healthy liver) and clinical outcomes in terms of toxicity and efficacy (i.e. radiological response).
Assessment of dosimetry and biodistribution based on quantitative assessment of imaging scans | 5 years
  Correlation between scout-based simulated absorbed dose (into the tumor and healthy liver) and the treatment based absorbed dose (into the tumor and healthy liver).
Quality of Life using EQ-5D-5L questionnaire | 1 year
  Patient reported outcome using EQ-5D-5L questionnaire. The scale measures quality of life on a 5-component scale including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.

CONTACTS AND LOCATIONS:
Overall Officials: Jens Ricke, Prof. Dr. med, Principal Investigator — Ludwig-Maximilian-University Munich (LMU); Wolfgang Weber, Prof. Dr. med, Principal Investigator — Munich Technische Universität (TUM); Thomas Kröncke, Prof. Dr. med, Principal Investigator — Universitätsklinikum Augsburg; Ralph Kickuth, Prof. Dr. med, Principal Investigator — Wuerzburg University Hospital; Karin Menhart, Dr., Principal Investigator — Universitätsklinikum Regensburg; Peter Dietrich, PD. Dr. med., Principal Investigator — Uniklinikum Erlangen
Locations (2):
- Germany (2):
  - Universitätsklinikum Augsburg, Augsburg
  - LMU Klinikum, Munich

IPD SHARING:
Plan to Share IPD: No